CLINICAL TRIAL: NCT02146456
Title: The Effect of Tranexamic Acid on Blood Coagulation After Colloid Infusion During Surgery: Rotational Thromboelastography Measurement
Brief Title: Rotational Thromboelastography Study in Tranexamic Acid and Colloid Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Pf, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Colloid_tranexamic acid
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Avascular Necrosis of Femoral Head; Degenerative Arthritis of Hip
MeSH Terms: conditions — Femur Head Necrosis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Colloid (No Intervention): During the operation, Lactate Ringer's solution is used as the maintenance fluid, and colloid is infused for the compensation of the intraoperative blood loss.
- Tranexamic acid (Experimental): During the operation, Lactate Ringer's solution is used as the maintenance fluid, and colloid is infused for the compensation of the intraoperative blood loss.
  In addition, 1 g of tranexamic acid in 100 ml normal saline is administered intravenously over 30 min after finishing the procedure of hip implant insertion.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid

SUMMARY:
Colloid solution is generally used to maintain intravascular volume. It is reported to impair blood coagulation in vivo and in vitro more than crystalloid does by prolonging coagulation time and decreasing clot strength. The formed fibrin clot is more vulnerable for fibrinolysis in a case of using colloid. Dilution of plasmin in vitro with colloid enhances fibrinolysis primarily by diminishing α2-antiplasmin-plasmin interaction.

Tranexamic acid is an antifibrinolytics that competitively inhibits the activation of plasminogen, by binding to specific site of both plasminogen and plasmin, a molecule responsible for the degradation of fibrin, a protein that forms the framework of blood clot. It is used to treat or prevent excessive blood loss during surgery and in other medical conditions. Gastrointestinal effect, dizziness, fatigue, headache, hypersensitivity reaction, or potential risk of thrombosis is reported as the adverse effect of tranexamic acid.

We hypothesized that inhibition of plasmin by tranexamic acid after colloid administration can improve the colloid-induced clot strength impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip replacement arthroplasty, who are diagnosed with the avascular necrosis of femoral head or degenerative arthritis of hip
* American Society of Anesthesiologist I or II

Exclusion Criteria:

* Patients receiving an intraoperative transfusion
* Patients receiving thrombin
* Patients having venous thromboembolism
* Patients having renal or hepatic disease
* Patients having coagulopathy
* Patient having heart failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Rotational thromboelastography | 30 minutes before starting an operation and 30 minutes after finishing an operation

SECONDARY OUTCOMES:
Hemoglobin | 30 minutes before starting an operation and 30 minutes after finishing an operation
Platelet | 30 minutes before starting an operation and 30 minutes after finishing an operation
International normalized ratio of prothrombin time | 30 minutes before starting an operation and 30 minutes after finishing an operation
Activated partial thromboplastin time | 30 minutes before starting an operation and 30 minutes after finishing an operation
Fibrinogen | 30 minutes before starting an operation and 30 minutes after finishing an operation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea